CLINICAL TRIAL: NCT07028970
Title: Long-term Follow-up Registry Study of Equecabtagene Autoleucel Injection
Status: Recruiting | Type: Observational
Sponsor: Nanjing IASO Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CT103AC003
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
Keywords: Long term follow up;; Eque-cel
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients received Equecabtagene Autoleucel Injection
  Interventions: Other: No Intervention (subjects were previously treated with Equecabtagene Autoleucel Injection) )

INTERVENTIONS:
Other: No Intervention (subjects were previously treated with Equecabtagene Autoleucel Injection) ) — This study is observational study and all participants will be obsreved with no intervention.

SUMMARY:
This is a multicenter, open-label, single-arm, long-term follow-up clinical study. All patients who have received Equecabtagene Autoleucel Injection treatment will be enrolled.

DETAILED DESCRIPTION:
The main follow-up period for pre-marketing clinical studies related to Equecabtagene Autoleucel Injection is 2 years. The "Technical Guidelines for Long-term Follow-up Clinical Studies of Gene Therapy Products (Trial)" issued by the Center for Drug Evaluation (CDE) of the National Medical Products Administration (NMPA) recommends a follow-up period of not less than 15 years for gene therapy products with genomic integration activity.

In order to observe the long-term safety and efficacy of Equecabtagene Autoleucel Injection, as well as the persistence of CAR-T cells in vivo, and to identify whether there are differences in safety among populations with different indications, this study will conduct long-term follow-up in patients treated with Equecabtagene Autoleucel Injection, thereby identifying long-term risks and helping to evaluate the product's benefit-risk profile.

ELIGIBILITY:
Inclusion Criteria:

- 1.Received Equecabtagene Autoleucel Injection treatment; 2.For those who participated in pre-marketing clinical studies or post-marketing real-world studies, must have completed or withdrawn from the original study; 3.Voluntary signing of an informed consent form approved by the ethics committee.

Exclusion Criteria:

* 1. Receipt of another lentiviral vector-based cell or gene therapy (either commercialized product or investigational product in a clinical tiral) between the infution of Equecabtagene Autoleucel Injection and the signing informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have received Equecabtagene Autoleucel Injection treatment. Patients who participated in pre-marketing clinical studies or post-marketing real-world studies with this product can only be enrolled after completing or prematurely withdrawing from their original studies.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2040-12 (Estimated); Study Completion 2043-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety profile of Equecabtagene Autoleucel Injection in treated patients. | Up to 15 years from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, PhD, Principal Investigator — Peking Union Medical College Hospital; Juan Du, PhD, Principal Investigator — RenJi Hospital
Locations (6):
- China (6):
  - Peking University First Hospital, Beijing
  - People's Hospital of Peking Universit, Beijing
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Henan Cancer Hospital Affilated Cancer Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No